CLINICAL TRIAL: NCT02556801
Title: A Single-center, Randomized, Double Blind, Placebo-Controlled, Parallel Group Study to Investigate the Relative Efficacy and Safety of Immunotherapy With SUBLIVAC FIX Phleum Pratense in Grass Pollen-Allergic Subjects With IgE-Mediated Seasonal ARC
Brief Title: Efficacy and Safety of SUBLIVAC Phleum for Immunotherapy of Grass Pollen-Allergy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HAL Allergy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP/0047
Record Dates: First submitted 2015-08-31; First posted 2015-09-22 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-08

CONDITIONS: Allergic Rhinitis; Allergic Rhinoconjunctivitis
Keywords: Sublingual immunotherapy; Dose range finding; Grass pollen; Allergic rhinitis/rhinoconjunctivitis; Immunogenicity
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind study
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SUBLIVAC FIX Phleum Prat. 0 AUN/ml (Placebo Comparator): 42 subjects received placebo (SUBLIVAC FIX Phleum Pratense 0 AUN/ml) sublingually. Subjects will start with one drop and add one drop each consecutive day until the maintenance dose of 5 drops per day is reached. Next treatment at maintenance dose is continued during 10 months.
  Interventions: Biological: SUBLIVAC FIX Phleum Prat.
- SUBLIVAC FIX Phleum Prat. 10,000 AUN/ml (Experimental): 42 subjects received SUBLIVAC FIX Phleum Pratense 10,000 AUN/ml) sublingually. Subjects will start with one drop and add one drop each consecutive day until the maintenance dose of 5 drops per day is reached. Next treatment at maintenance dose is continued during 10 months.
  Interventions: Biological: SUBLIVAC FIX Phleum Prat.
- SUBLIVAC FIX Phleum Prat. 40,000 AUN/ml (Experimental): 40 subjects received SUBLIVAC FIX Phleum Pratense 40,000 AUN/ml sublingually. Subjects will start with one drop and add one drop each consecutive day until the maintenance dose of 5 drops per day is reached. Next treatment at maintenance dose is continued during 10 months.
  Interventions: Biological: SUBLIVAC FIX Phleum Prat.
- SUBLIVAC FIX Phleum Prat. 80,000 AUN/ml (Experimental): 40 subjects received SUBLIVAC FIX Phleum Pratense 80,000 AUN/ml sublingually. Subjects will start with one drop and add one drop each consecutive day until the maintenance dose of 5 drops per day is reached. Next treatment at maintenance dose is continued during 10 months.
  Interventions: Biological: SUBLIVAC FIX Phleum Prat.

INTERVENTIONS:
Biological: SUBLIVAC FIX Phleum Prat. — sublingual daily administration

SUMMARY:
The purpose of this study is to assess safety, tolerability and demonstrate a dose response signal using Total Symptom Score (TSS), based on challenges with grass pollen in an Environmental Exposure Chamber (EEC), followed by estimation of the minimum effective dose of SUBLIVAC FIX Phleum (SP) after 10 months of treatment compared to placebo.

The study has 4 treatment groups: 3 different doses of SP and placebo will be tested.

DETAILED DESCRIPTION:
The current dose range finding study with SP has been designed to test three different concentrations of SUBLIVAC FIX Phleum (SP) that includes 3 doses (10,000 AUN/mL; 40,000 AUN/mL; 80,000 AUN/mL) and placebo to demonstrate a dose response signal and to estimate the minimal effective dose of SP. The study will be conducted in the target population of seasonal allergic subjects in a fully validated Environmental Exposure Chamber (EEC) system. The EEC system is a facility that has temporal uniformity of airborne allergen (pollen) exposure to subjects. Use of the EEC ensures exposure to relatively consistent levels of allergen. This facility has been used in a number of immunotherapy trials and is an improved challenge model of AR compared to the previously used nasal provocation test. Treatment duration of this study is extended to 10 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who signed informed consent.
2. Subjects aged ≥18 and ≤65 years at signing of informed consent.
3. Subjects with at least two-year clinical history of allergic rhinitis/rhinoconjunctivitis to grass pollen, with or without concomitant asthma (asthma must be controlled).
4. Subjects with a forced expiratory volume at one second (FEV1) >70% of the predicted value as measured during screening or documented within 1 year of study start.
5. Subjects with a positive skin prick test (SPT) (mean wheal diameter of at least 3 mm larger than the negative control; negative control should be <2 mm, histamine control should be positive (mean wheal diameter of at least 3 mm larger than the negative control)) for grass pollen assessed during screening or a documented positive response obtained within 1 year before screening.
6. Subjects with a grass pollen specific IgE greater than or equal to 0.7 kiloUnits (kU)/L assessed during screening or a documented positive result obtained within 1 year before screening.
7. Subjects with a TSS of at least 10/24 during baseline EEC challenge (V2) in combination with a staff assessed score of at least 2/3 for two objective TSS symptoms (i.e. running nose, sneezing or red eyes), during the baseline EEC challenge.

Exclusion Criteria:

1. Subjects with (expected) clinically relevant symptoms at the timing of the scheduled EEC assessments at Visit 2 and Visit 6 due to concomitant sensitization i.e. positive SPT (mean wheal diameter of at least 3 mm larger than the negative control) and a history of allergic response to the causative allergen, at the discretion of the investigator.
2. Patients with grass pollen induced asthma.
3. Subjects who cannot tolerate the Baseline Challenge in the EEC.
4. Subjects who received immunotherapy (SCIT or SLIT) with grass pollen allergens within the past 5 years.
5. (Ongoing) allergen-specific immunotherapy with any allergen(s) during the study period.
6. Subjects with unsuccessful allergen-specific immunotherapy within the past 5 years (e.g., but not limited to, prematurely stopped immunotherapy due to non-compliance, AEs or lack of therapeutic effect), at the discretion of the investigator.
7. Subjects undergoing anti-IgE therapy within the 6 months prior to inclusion and/or during the study.
8. Subjects suffering from severe immune disorders (including auto-immune diseases) and/or diseases requiring immunosuppressive drugs.
9. Subjects suffering from active malignancies or any malignant disease (except for localized basal cell cancers of the skin as long as they have been adequately treated and no recurrence within 3 months of screening visit) during 5 years prior to screening.
10. Subjects suffering from severe uncontrolled diseases that could increase the risk for participating in the study, including but not limited to: cardiovascular insufficiency, any severe or unstable lung diseases, endocrine diseases, clinically significant renal or hepatic diseases, or haematological disorders at the discretion of the Investigator.
11. Subjects who have active inflammation or infection of the target organs (nose, eyes or lower airways) at Visit 1.
12. Subjects suffering from diseases with a contraindication for the use of adrenaline (e.g. hyperthyroidism, glaucoma).
13. Subjects receiving vaccination within one week before start of therapy or during the up-dosing phase.
14. Subjects receiving treatment with systemic steroids within 4 weeks before visit 1 and/or during the study.
15. Subjects receiving treatment with systemic or local β-blockers anytime during the study.
16. Subjects who participated in a clinical study within the last 3 months (e.g. new investigational drug or biological) or within the last 30 days (e.g. bio-equivalent drug), at the discretion of the Investigator.
17. Female subjects of child-bearing potential who are pregnant, lactating or using inadequate contraceptive measures (adequate contraceptive measures will be: sexual abstinence; oral contraceptives, trans dermal patches or depot injection of a progestogen drug (starting at least 4 weeks prior to investigational medicinal product (IMP) administration); double barrier method: condom or occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent; intrauterine device (IUD), intrauterine system (IUS), implant, or vaginal ring (placed at least 4 weeks prior to IMP administration); or male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into trial and is the sole sexual partner for that female subject.
18. Subjects that have a history of alcohol, drug or medication abuse within the past year before study start.
19. Subjects with any clinically relevant abnormal laboratory parameter at screening.
20. Subjects that lack cooperation or compliance, as judged by the investigator.
21. Subjects suffering from severe psychiatric, psychological, or neurological disorders.
22. Subjects who are employees of the sponsor or contract research organisation and/or 1st grade relatives or partners of the (principal) investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Couroux, MD, Principal Investigator — Inflamax
Locations (1):
- Inflamax Research Inc., Mississauga, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The total recruitment period of the study was from September until November 2015. As soon as approx. 160 subjects had been randomized, recruitment was stopped and the investigator was informed to end recruitment of patients. Already screened patients were randomized, if eligible. See summary in the table below.
Groups:
- Placebo: Subjects received placebo (containing no allergen extract) sublingually. Subjects started with one drop and one drop was added each consecutive day until the maintenance dose of 5 drops per day was reached. Next treatment at maintenance dose was continued during 10 months.
- SP 10,000 AUN/ml: Subjects received SUBLIVAC FIX Phleum Pratense 10,000 AUN/ml) sublingually. Subjects started with one drop and one drop was added each consecutive day until the maintenance dose of 5 drops per day was reached. Next treatment at maintenance dose was continued during 10 months.
- SP 40,000 AUN/ml: Subjects received SUBLIVAC FIX Phleum Pratense 40,000 AUN/ml sublingually. Subjects started with one drop and one drop was added each consecutive day until the maintenance dose of 5 drops per day was reached. Next treatment at maintenance dose was continued during 10 months.
- SP 80,000 AUN/ml: Subjects received SUBLIVAC FIX Phleum Pratense 80,000 AUN/ml sublingually. Subjects started with one drop and one drop was added each consecutive day until the maintenance dose of 5 drops per day was reached. Next treatment at maintenance dose was continued during 10 months.
Period: Overall Study
Arm/Group | Placebo | SP 10,000 AUN/ml | SP 40,000 AUN/ml | SP 80,000 AUN/ml
Started | 42 | 42 | 42 | 42
Completed | 40 | 35 | 38 | 37
Not Completed | 2 | 7 | 4 | 5
Not completed — Lost to Follow-up | 1 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 3 | 1 | 1
Not completed — Adverse Event | 0 | 2 | 0 | 3
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Personal reasons patient | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Patients received placebo (containing no allergen extract) sublingually. Subjects started with one drop and one drop was added each consecutive day until the maintenance dose of 5 drops per day was reached. Next treatment at maintenance dose was continued during 10 months.
- SP 10,000 AUN/ml: Patients received SUBLIVAC FIX Phleum Pratense 10,000 AUN/ml) sublingually. Subjects started with one drop and one drop was added each consecutive day until the maintenance dose of 5 drops per day was reached. Next treatment at maintenance dose was continued during 10 months.
- SP 40,000 AUN/ml: Patients received SUBLIVAC FIX Phleum Pratense 40,000 AUN/ml sublingually. Subjects started with one drop and one drop was added each consecutive day until the maintenance dose of 5 drops per day was reached. Next treatment at maintenance dose was continued during 10 months.
- SP 80,000 AUN/ml: Patients received SUBLIVAC FIX Phleum Pratense 80,000 AUN/ml sublingually. Subjects started with one drop and one drop was added each consecutive day until the maintenance dose of 5 drops per day was reached. Next treatment at maintenance dose was continued during 10 months.
- Total: Total of all reporting groups
Arm/Group | Placebo | SP 10,000 AUN/ml | SP 40,000 AUN/ml | SP 80,000 AUN/ml | Total
Number analyzed (Participants) | 42 | 42 | 42 | 42 | 168
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 0 | 1
  Between 18 and 65 years | 41 | 42 | 42 | 42 | 167
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (12.1) | 42.4 (11.6) | 39.2 (10.6) | 40.9 (10.4) | 40.5 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 23 | 22 | 28 | 100
  Male | 15 | 19 | 20 | 14 | 68
Region of Enrollment [Number; unit: participants]
  Canada | 42 | 42 | 42 | 42 | 168

OUTCOME MEASURES:

1. Primary Outcome: Mean Total Symptom Score (TSS) After 10 Months of Treatment (Visit 6) Compared to Placebo
Description: The primary endpoint was the TSS after 10 months of treatment (at visit 6). The mean TSS at visit 6 was calculated as an average of all non-missing TSS scores between 1 and 6 hours after start of Environmental Exposure Chamber (EEC) challenge at visit 6. TSS was computed as the sum of individual scores for eight nasal and non-nasal symptoms (rhinorrhea, congestion, sneezing, itchiness, itchy/gritty eyes, tearing/watery eyes, red/burning eyes, and ear/palate itching). Each of eight symptoms was rated on a scale of 0-3 as follows: 0, none; 1, mild; 2, moderate; 3, severe. The range of TSS is from 0 to 24 units on a scale. The highest the score, the more severe symptoms a subject experiences. Negative change of TSS between baseline and visit 6 was expected (reduced symptoms), more negative change at visit 6 versus baseline represents better outcome of the study.
Time Frame: 10 months after treatment start (baseline - Visit 2)
Population: The Intention-to-Treat population (ITT) includes all randomized subjects who received at least one dose of the study drug and for whom at least one post-baseline measurement for the primary efficacy endpoint was available.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | SP 10,000 AUN/ml | SP 40,000 AUN/ml | SP 80,000 AUN/ml
Number analyzed (Participants) | 40 | 35 | 38 | 37
Score on a scale | 10.01 (0.80) | 8.06 (0.85) | 8.19 (0.82) | 7.69 (0.83)
Statistical Analysis 1: Comparison: Placebo vs SP 10,000 AUN/ml vs SP 40,000 AUN/ml vs SP 80,000 AUN/ml; Test type: Superiority; p = 0.057, MCP-Mod Method; The primary dose-response analysis was performed by applying linear, Emax, logistic and exponential models.The p-value was based on Emax model; Test statistic = 1.823
Statistical Analysis 2: Comparison: Placebo vs SP 10,000 AUN/ml; Test type: Superiority; Treatment effect = -1.96, 90% CI 2-sided [-3.89 to -0.03], Standard Deviation 1.17
Statistical Analysis 3: Comparison: Placebo vs SP 40,000 AUN/ml; Test type: Superiority; Treatment effect = -1.83, 90% CI 2-sided [-3.72 to 0.06], Standard Error of Mean 1.14
Statistical Analysis 4: Comparison: Placebo vs SP 80,000 AUN/ml; Test type: Superiority; Treatment effect = -2.33, 90% CI 2-sided [-4.23 to -0.43], Standard Error of Mean 1.15

2. Secondary Outcome: Change From Baseline in Mean Total Symptom Score (TSS) After 10 Months of Treatment (Visit 6)
Description: The change from baseline of the mean TSS at visit 6. The baseline will be calculated as an average of all non-missing TSS scores between 1 and 6 hours after start of Environmental Exposure Chamber (EEC) challenge at visit 2. The range of TSS is from 0 to 24 units on a scale. The highest the score, the more severe symptoms a subject experiences. Negative change of TSS between baseline and visit 6 was expected (reduced symptoms), more negative change at visit 6 versus baseline represents better outcome of the study.
Time Frame: 10 months after treatment start compared to first day of treatment (TSS at baseline measured at Visit 2, before IMP administration)
Population: The Intention-to-Treat population (ITT) consists of all randomized subjects who received at least one dose of the study drug and for whom at least one post-baseline measurement for the primary efficacy endpoint was available.
Measure: Least Squares Mean (Standard Error); unit: mean Total Symptom Score
Arm/Group | Placebo | SP 10,000 AUN/ml | SP 40,000 AUN/ml | SP 80,000 AUN/ml
Number analyzed (Participants) | 40 | 35 | 38 | 37
mean Total Symptom Score | -3.45 (0.80) | -5.37 (0.85) | -5.24 (0.81) | -5.74 (0.83)
Statistical Analysis 1: Comparison: Placebo vs SP 10,000 AUN/ml; Test type: Superiority; p = 0.051, Mixed Models Analysis; Treatment effect = -1.92, 90% CI 2-sided [-3.85 to 0.01], Standard Error of Mean 1.17
Statistical Analysis 2: Comparison: Placebo vs SP 40,000 AUN/ml; Test type: Superiority; p = 0.059, Mixed Models Analysis; Treatment effect = -1.79, 90% CI 2-sided [-3.68 to 0.10], Standard Error of Mean 1.14
Statistical Analysis 3: Comparison: Placebo vs SP 80,000 AUN/ml; Test type: Superiority; p = 0.024, Mixed Models Analysis; Treatment effect = -2.30, 90% CI 2-sided [-4.20 to -0.40], Standard Error of Mean 1.15

3. Secondary Outcome: Change From Baseline in Mean Total Symptom Score (TSS) After 5 Months of Treatment (Visit 4)
Description: The change from baseline of the mean TSS at visit 4. The mean TSS at visit 4 will be calculated as an average of all non-missing TSS between 1 and 6 hours after start of Environmental Exposure Chamber (EEC) challenge at visit 4. The baseline will be calculated as an average of all non-missing TSS between 1 and 6 hours after start of EEC challenge at visit 2. The range of TSS is from 0 to 24 units on a scale. The highest the score, the more severe symptoms a subject experiences. Negative change of TSS between baseline and visit 4 was expected (reduced symptoms), more negative change at visit 4 versus baseline represents better outcome of the study.The highest the score, the more severe symptoms a subject experiences.
Time Frame: 5 months after treatment start compared to first day of treatment (TSS at baseline measured at Visit 2, before IMP administration)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mean Total Symptom Score
Arm/Group | Placebo | SP 10,000 AUN/ml | SP 40,000 AUN/ml | SP 80,000 AUN/ml
Number analyzed (Participants) | 40 | 35 | 38 | 37
mean Total Symptom Score | -2.40 (0.74) | -3.00 (0.79) | -4.24 (0.76) | -4.18 (0.78)
Statistical Analysis 1: Comparison: Placebo vs SP 10,000 AUN/ml; Test type: Superiority; p = 0.291, Mixed Models Analysis; Treatment effect = -0.60, 90% CI 2-sided [-2.39 to 1.19], Standard Error of Mean 1.08
Statistical Analysis 2: Comparison: Placebo vs SP 40,000 AUN/ml; Test type: Superiority; p = 0.042, Mixed Models Analysis; Treatment effect = -1.84, 90% CI 2-sided [-3.60 to -0.09], Standard Error of Mean 1.06
Statistical Analysis 3: Comparison: Placebo vs SP 80,000 AUN/ml; Test type: Superiority; p = 0.050, Mixed Models Analysis; Treatment effect = -1.78, 90% CI 2-sided [-3.56 to 0.00], Standard Error of Mean 1.08

4. Secondary Outcome: Change From Baseline in Mean Total Nasal Symptom Score (TNSS) After 10 Months of Treatment (Visit 6)
Description: The change from baseline of the mean TNSS at visit 6. The mean TNSS at visit 6 will be calculated as an average of all non-missing TNSS between 1 and 6 hours after start of EEC challenge at visit 6. The baseline will be calculated as an average of all non-missing TNSS between 1 and 6 hours after start of Environmental Exposure Chamber (EEC) challenge at visit 2. TNSS will be computed as the sum of individual scores for four nasal symptoms (running nose, congestion, itchy nose, and sneezing). Each of the four symptoms will be rated on a scale of 0-3 as follows: 0, none; 1, mild; 2, moderate; and 3, severe. The range of TNSS is from 0 to 12 units on a scale. The highest the score, the more severe symptoms a subject experiences.Negative change of TNSS between baseline and visit 6 was expected (reduced symptoms), more negative change at visit 6 versus baseline represents better outcome of the study.
Time Frame: 10 months after treatment start compared to first day of treatment (TSS at baseline measured at Visit 2, before IMP injection)
Measure: Least Squares Mean (Standard Error); unit: mean Total Nasal Symptom Score
Arm/Group | Placebo | SP 10,000 AUN/ml | SP 40,000 AUN/ml | SP 80,000 AUN/ml
Number analyzed (Participants) | 40 | 35 | 38 | 37
mean Total Nasal Symptom Score | -1.87 (0.43) | -2.76 (0.46) | -2.75 (0.44) | -2.98 (0.44)
Statistical Analysis 1: Comparison: Placebo vs SP 10,000 AUN/ml; Test type: Superiority; p = 0.079, Mixed Models Analysis; Treatment effect = -0.89, 90% CI 2-sided [-1.93 to 0.15], Standard Error of Mean 0.63
Statistical Analysis 2: Comparison: Placebo vs SP 40,000 AUN/ml; Test type: Superiority; p = 0.076, Mixed Models Analysis; Treatment effect = -0.88, 90% CI 2-sided [-1.89 to 0.13], Standard Error of Mean 0.61
Statistical Analysis 3: Comparison: Placebo vs SP 80,000 AUN/ml; Test type: Superiority; p = 0.038, Mixed Models Analysis; Treatment effect = -1.11, 0.62% CI 2-sided [-2.13 to -0.08], Standard Error of Mean 0.62

5. Secondary Outcome: Change From Baseline in Mean Total Nasal Symptom Score (TNSS) After 5 Months of Treatment (Visit 4)
Description: The change from baseline of the mean TNSS at visit 4. The mean TNSS at visit 4 will be calculated as an average of all non-missing TNSS between 1 and 6 hours after start of Environmental Exposure Chamber (EEC) challenge at visit 4. The baseline will be calculated as an average of all non-missing TNSS between 1 and 6 hours after start of during EEC challenge at visit 2. TNSS will be computed as the sum of individual scores for four nasal symptoms (running nose, congestion, itchy nose, and sneezing). Each of the four symptoms will be rated on a scale of 0-3 as follows: 0, none; 1, mild; 2, moderate; and 3, severe. The range of TNSS is from 0 to 12 units on a scale. The highest the score, the more severe symptoms a subject experiences. Negative change of TSS between baseline and visit 6 was expected (reduced symptoms), more negative change at visit 4 versus baseline represents better outcome of the study.
Time Frame: 5 months after treatment start compared to first day of treatment (TSS at baseline measured at Visit 2, before IMP injection)
Measure: Least Squares Mean (Standard Error); unit: mean Total Nasal Symptom Score
Arm/Group | Placebo | SP 10,000 AUN/ml | SP 40,000 AUN/ml | SP 80,000 AUN/ml
Number analyzed (Participants) | 40 | 35 | 38 | 37
mean Total Nasal Symptom Score | -1.52 (0.39) | -1.59 (0.42) | -2.14 (0.40) | -2.02 (0.42)
Statistical Analysis 1: Comparison: Placebo vs SP 10,000 AUN/ml; Test type: Superiority; p = 0.451, Mixed Models Analysis; Treatment effect = -0.07, 90% CI 2-sided [-1.03 to 0.88], Standard Error of Mean 0.58
Statistical Analysis 2: Comparison: Placebo vs SP 40,000 AUN/ml; Test type: Superiority; p = 0.137, Mixed Models Analysis; Treatment effect = -0.62, 90% CI 2-sided [-1.55 to 0.32], Standard Error of Mean 0.56
Statistical Analysis 3: Comparison: Placebo vs SP 80,000 AUN/ml; Test type: Superiority; p = 0.195, Mixed Models Analysis; Treatment effect = -0.500, 90% CI 2-sided [-1.45 to 0.46], Standard Error of Mean 0.57

6. Secondary Outcome: Mean Combined Symptom and Medication Scores (CSMS) During the Grass Pollen Season.
Description: The mean CSMS will be calculated as an average of all non-missing daily CSMS during the grass pollen season. Subjects that did not complete at least 75% of their diary data, and subjects who have been on holidays outside the region for more than 7 days during the actual grass pollen season will be excluded from the analysis. The daily CSMS will be computed according to the definition given by the EAACI Position Paper. The actual grass pollen season would start on the first of 3 consecutive days that have a grass pollen count ≥ 10 ppm3 per 24 hours and the season would end on the first of 3 consecutive days that have a grass pollen count < 10 ppm3 per 24 hours. The defined pollen season could consist of several separate periods that comply with this definition. The CSMS has a range from 0 to 6 and the higher the score, the more severe symptoms a subject is experiencing.
Time Frame: during the grass pollen season: estimated between 6 and 10 months after start of treatment at Visit 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mean Combined Symptom Medication Score
Arm/Group | Placebo | SP 10,000 AUN/ml | SP 40,000 AUN/ml | SP 80,000 AUN/ml
Number analyzed (Participants) | 40 | 35 | 38 | 37
mean Combined Symptom Medication Score | 1.032 (0.135) | 0.678 (0.124) | 0.638 (0.128) | 0.752 (0.122)
Statistical Analysis 1: Comparison: Placebo vs SP 10,000 AUN/ml; Test type: Superiority; p = 0.028, ANOVA; Treatment effect = -0.354, 90% CI 2-sided [-0.657 to -0.050], Standard Error of Mean 0.183
Statistical Analysis 2: Comparison: Placebo vs SP 40,000 AUN/ml; Test type: Superiority; p = 0.018, ANOVA; Treatment effect = -0.394, 90% CI 2-sided [-0.702 to -0.086], Standard Error of Mean 0.186
Statistical Analysis 3: Comparison: Placebo vs SP 80,000 AUN/ml; Test type: Superiority; p = 0.063, ANOVA; Treatment effect = -0.280, 90% CI 2-sided [-0.581 to 0.021], Standard Error of Mean 0.182

7. Secondary Outcome: Change From Baseline in Serum Specific Immunoglobulin (IgE) Levels After 5 Months (Visit 4) and 10 Months (Visit 6) of Treatment
Description: Changes from baseline in serum specific immunoglobulin levels (IgE) after after 5 months of treatment (Visit 4) and after 10 months of treatment (Visit 6). Measurements at visit 1 will be used as baseline.
Time Frame: 5 and 10 months after treatment start compared to first day of treatment (IgE at baseline measured at Visit 2, before IMP administration)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean fold change
Arm/Group | Placebo | SP 10,000 AUN/ml | SP 40,000 AUN/ml | SP 80,000 AUN/ml
Number analyzed (Participants) | 40 | 35 | 38 | 37
Geometric Mean fold change
  After 5 months (Visit 4) | 1.48 [1.15 to 1.89] | 2.83 [2.17 to 3.69] | 3.59 [2.78 to 4.62] | 3.45 [2.67 to 4.46]
  After 10 months (Visit 6) | 1.73 [1.35 to 2.22] | 2.47 [1.89 to 3.22] | 2.90 [2.25 to 3.73] | 2.37 [1.84 to 3.07]
Statistical Analysis 1: Comparison: Placebo vs SP 10,000 AUN/ml; Analysis of change from baseline of serum specific IgE levels after 5 months (Visit 4); Test type: Superiority; p < 0.001, Mixed Models Analysis; Treatment effect = 1.92, 90% CI 2-sided [1.41 to 2.60]
Statistical Analysis 2: Comparison: Placebo vs SP 40,000 AUN/ml; Analysis of change from baseline of serum specific IgE levels after 5 months (Visit 4); Test type: Superiority; p < 0.001, Mixed Models Analysis; Treatment effect = 2.43, 90% CI 2-sided [1.80 to 3.27]
Statistical Analysis 3: Comparison: Placebo vs SP 80,000 AUN/ml; Analysis of change from baseline of serum specific IgE levels after 5 months (Visit 4); Test type: Superiority; p < 0.001, Mixed Models Analysis; Treatment effect = 2.34, 90% CI 2-sided [1.73 to 3.15]
Statistical Analysis 4: Comparison: Placebo vs SP 10,000 AUN/ml; Analysis of change from baseline of serum specific IgE levels after 10 months (Visit 6); Test type: Superiority; p = 0.029, Mixed Models Analysis; Treatment effect = 1.42, 90% CI 2-sided [1.05 to 1.93]
Statistical Analysis 5: Comparison: Placebo vs SP 40,000 AUN/ml; Analysis of change from baseline of serum specific IgE levels after 10 months (Visit 6); Test type: Superiority; p = 0.003, Mixed Models Analysis; Treatment effect = 1.67, 90% CI 2-sided [1.24 to 2.25]
Statistical Analysis 6: Comparison: Placebo vs SP 80,000 AUN/ml; Analysis of change from baseline of serum specific IgE levels after 10 months (Visit 6); Test type: Superiority; p = 0.042, Mixed Models Analysis; Treatment effect = 1.37, 90% CI 2-sided [1.01 to 1.85]

8. Secondary Outcome: Change From Baseline in Serum Specific Immunoglobulin (IgG) Levels After 5 Months (Visit 4) and 10 Months (Visit 6) of Treatment
Description: Changes from baseline in serum specific immunoglobulin levels (IgG ATG, IgG AP1 and IgG AP5) after after 5 months of treatment (Visit 4) and after 10 months of treatment (Visit 6). Measurements at visit 1 will be used as baseline.
Time Frame: 5 and 10 months after treatment start compared to first day of treatment (IgG at baseline measured at Visit 2, before IMP injection)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean fold change
Arm/Group | Placebo | SP 10,000 AUN/ml | SP 40,000 AUN/ml | SP 80,000 AUN/ml
Number analyzed (Participants) | 40 | 35 | 38 | 37
Geometric Mean fold change
  IgG ATG after 5 months (Visit 4) | 0.99 [0.91 to 1.08] | 1.10 [1.00 to 1.20] | 1.28 [1.18 to 1.40] | 1.23 [1.13 to 1.34]
  IgG ATG after 10 months (Visit 6) | 0.98 [0.86 to 1.11] | 1.21 [1.05 to 1.39] | 1.57 [1.37 to 1.79] | 1.36 [1.19 to 1.55]
  IgG AP1 after 5 months (Visit 4) | 0.98 [0.94 to 1.03] | 0.97 [0.92 to 1.02] | 1.08 [1.03 to 1.13] | 1.00 [0.96 to 1.05]
  IgG AP1 after 10 months (Visit 6) | 0.99 [0.93 to 1.05] | 1.01 [0.94 to 1.07] | 1.20 [1.13 to 1.28] | 1.10 [1.03 to 1.17]
  IgG AP5 after 5 months (Visit 4) | 0.99 [0.92 to 1.06] | 1.03 [0.96 to 1.11] | 1.15 [1.07 to 1.24] | 1.14 [1.06 to 1.22]
  IgG AP5 after 10 months (Visit 6) | 0.98 [0.88 to 1.09] | 1.07 [0.96 to 1.20] | 1.25 [1.12 to 1.39] | 1.23 [1.11 to 1.37]
Statistical Analysis 1: Comparison: Placebo vs SP 10,000 AUN/ml; Analysis of change from baseline of serum specific IgG ATG levels after 5 months (Visit 4); Test type: Superiority; p = 0.057, Mixed Models Analysis; Treatment effect = 1.11, 90% CI 2-sided [1.00 to 1.23]
Statistical Analysis 2: Comparison: Placebo vs SP 40,000 AUN/ml; Analysis of change from baseline of serum specific IgG ATG levels after 5 months (Visit 4); Test type: Superiority; p < 0.001, Mixed Models Analysis; Treatment effect = 1.29, 90% CI 2-sided [1.17 to 1.43]
Statistical Analysis 3: Comparison: Placebo vs SP 80,000 AUN/ml; Analysis of change from baseline of serum specific IgG ATG levels after 5 months (Visit 4); Test type: Superiority; p < 0.001, Mixed Models Analysis; Treatment effect = 1.24, 90% CI 2-sided [1.12 to 1.37]
Statistical Analysis 4: Comparison: Placebo vs SP 10,000 AUN/ml; Analysis of change from baseline of serum specific IgG ATG levels after 10 months (Visit 6); Test type: Superiority; p = 0.015, Mixed Models Analysis; Treatment effect = 1.23, 90% CI 2-sided [1.05 to 1.45]
Statistical Analysis 5: Comparison: Placebo vs SP 40,000 AUN/ml; Analysis of change from baseline of serum specific IgG ATG levels after 10 months (Visit 6); Test type: Superiority; p < 0.001, Mixed Models Analysis; Treatment effect = 1.60, 90% CI 2-sided [1.37 to 1.87]
Statistical Analysis 6: Comparison: Placebo vs SP 80,000 AUN/ml; Analysis of change from baseline of serum specific IgG ATG levels after 10 months (Visit 6); Test type: Superiority; p < 0.001, Mixed Models Analysis; Treatment effect = 1.39, 90% CI 2-sided [1.19 to 1.62]
Statistical Analysis 7: Comparison: Placebo vs SP 10,000 AUN/ml; Analysis of change from baseline of serum specific IgG AP1 levels after 5 months (Visit 4); Test type: Superiority; p = 0.341, Mixed Models Analysis; Treatment effect = 0.99, 90% CI 2-sided [0.93 to 1.04]
Statistical Analysis 8: Comparison: Placebo vs SP 40,000 AUN/ml; Analysis of change from baseline of serum specific IgG AP1 levels after 5 months (Visit 4); Test type: Superiority; p = 0.003, Mixed Models Analysis; Treatment effect = 1.10, 90% CI 2-sided [1.04 to 1.16]
Statistical Analysis 9: Comparison: Placebo vs SP 80,000 AUN/ml; Analysis of change from baseline of serum specific IgG AP1 levels after 5 months (Visit 4); Test type: Superiority; p = 0.269, Mixed Models Analysis; Treatment effect = 1.02, 90% CI 2-sided [0.97 to 1.08]
Statistical Analysis 10: Comparison: Placebo vs SP 10,000 AUN/ml; Analysis of change from baseline of serum specific IgG AP1 levels after 10 months (Visit 6); Test type: Superiority; p = 0.312, Mixed Models Analysis; Treatment effect = 1.02, 90% CI 2-sided [0.95 to 1.10]
Statistical Analysis 11: Comparison: Placebo vs SP 40,000 AUN/ml; Analysis of change from baseline of serum specific IgG AP1 levels after 10 months (Visit 6); Test type: Superiority; p < 0.001, Mixed Models Analysis; Treatment effect = 1.22, 90% CI 2-sided [1.13 to 1.31]
Statistical Analysis 12: Comparison: Placebo vs SP 80,000 AUN/ml; Analysis of change from baseline of serum specific IgG AP1 levels after 10 months (Visit 6); Test type: Superiority; p = 0.008, Mixed Models Analysis; Treatment effect = 1.11, 90% CI 2-sided [1.03 to 1.20]
Statistical Analysis 13: Comparison: Placebo vs SP 10,000 AUN/ml; Analysis of change from baseline of serum specific IgG AP5 levels after 5 months (Visit 4); Test type: Superiority; p = 0.212, Mixed Models Analysis; Treatment effect = 1.04, 90% CI 2-sided [0.96 to 1.14]
Statistical Analysis 14: Comparison: Placebo vs SP 40,000 AUN/ml; Analysis of change from baseline of serum specific IgG AP5 levels after 5 months (Visit 4); Test type: Superiority; p = 0.002, Mixed Models Analysis; Treatment effect = 1.16, 90% CI 2-sided [1.07 to 1.27]
Statistical Analysis 15: Comparison: Placebo vs SP 80,000 AUN/ml; Analysis of change from baseline of serum specific IgG AP5 levels after 5 months (Visit 4); Test type: Superiority; p = 0.004, Mixed Models Analysis; Treatment effect = 1.15, 90% CI 2-sided [1.06 to 1.25]
Statistical Analysis 16: Comparison: Placebo vs SP 10,000 AUN/ml; Analysis of change from baseline of serum specific IgG AP5 levels after 10 months (Visit 6); Test type: Superiority; p = 0.126, Mixed Models Analysis; Treatment effect = 1.09, 90% CI 2-sided [0.96 to 1.24]
Statistical Analysis 17: Comparison: Placebo vs SP 40,000 AUN/ml; Analysis of change from baseline of serum specific IgG AP5 levels after 10 months (Visit 6); Test type: Superiority; p < 0.001, Mixed Models Analysis; Treatment effect = 1.28, 90% CI 2-sided [1.13 to 1.45]
Statistical Analysis 18: Comparison: Placebo vs SP 80,000 AUN/ml; Analysis of change from baseline of serum specific IgG AP5 levels after 10 months (Visit 6); Test type: Superiority; p = 0.002, Mixed Models Analysis; Treatment effect = 1.26, 90% CI 2-sided [1.11 to 1.43]

9. Secondary Outcome: Change From Baseline in Serum Specific Immunoglobulin (IgG4) Levels After 5 Months (Visit 4) and 10 Months (Visit 6) of Treatment
Description: Changes from baseline in serum specific immunoglobulin levels (IgG4 ATG, IgG4 AP1 and IgG4 AP5) after 5 months of treatment (Visit 4) and after 10 months of treatment (Visit 6). Measurements at visit 1 will be used as baseline.
Time Frame: 5 and 10 months after treatment start compared to first day of treatment (IgG4 at baseline measured at Visit 2, before IMP injection)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean fold change
Arm/Group | Placebo | SP 10,000 AUN/ml | SP 40,000 AUN/ml | SP 80,000 AUN/ml
Number analyzed (Participants) | 40 | 35 | 38 | 37
Geometric Mean fold change
  IgG4 ATG after 5 months (Visit 4) | 1.01 [0.83 to 1.24] | 1.34 [1.08 to 1.67] | 2.18 [1.77 to 2.68] | 2.05 [1.67 to 2.54]
  IgG4 ATG after 10 months (Visit 6) | 1.11 [0.85 to 1.46] | 1.65 [1.24 to 2.20] | 3.21 [2.44 to 4.23] | 2.36 [1.79 to 3.12]
  IgG4 AP1 after 5 months (Visit 4) | 1.04 [0.87 to 1.24] | 1.22 [1.02 to 1.48] | 2.06 [1.72 to 2.47] | 1.63 [1.36 to 1.95]
  IgG4 AP1 after 10 months (Visit 6) | 1.12 [0.90 to 1.39] | 1.56 [1.24 to 1.96] | 2.66 [2.14 to 3.32] | 1.90 [1.52 to 2.37]
  IgG4 AP5 after 5 months (Visit 4) | 1.03 [0.73 to 1.44] | 1.57 [1.09 to 2.25] | 2.42 [1.71 to 3.42] | 2.91 [2.05 to 4.13]
  IgG5 AP5 after 10 months (Visit 6) | 1.16 [0.79 to 1.72] | 1.94 [1.28 to 2.94] | 3.12 [2.09 to 4.66] | 3.35 [2.23 to 5.03]
Statistical Analysis 1: Comparison: Placebo vs SP 10,000 AUN/ml; Analysis of change from baseline of serum specific IgG4 ATG levels after 5 months (Visit 4); Test type: Superiority; p = 0.032, Mixed Models Analysis; Treatment effect = 1.33, 90% CI 2-sided [1.03 to 1.70]
Statistical Analysis 2: Comparison: Placebo vs SP 40,000 AUN/ml; Analysis of change from baseline of serum specific IgG4 ATG levels after 5 months (Visit 4); Test type: Superiority; p < 0.001, Mixed Models Analysis; Treatment effect = 2.15, 90% CI 2-sided [1.68 to 2.74]
Statistical Analysis 3: Comparison: Placebo vs SP 80,000 AUN/ml; Analysis of change from baseline of serum specific IgG4 ATG levels after 5 months (Visit 4); Test type: Superiority; p < 0.001, Mixed Models Analysis; Treatment effect = 2.03, 90% CI 2-sided [1.59 to 2.59]
Statistical Analysis 4: Comparison: Placebo vs SP 10,000 AUN/ml; Analysis of change from baseline of serum specific IgG4 ATG levels after 10 months (Visit 6); Test type: Superiority; p = 0.024, Mixed Models Analysis; Treatment effect = 1.48, 90% CI 2-sided [1.07 to 2.06]
Statistical Analysis 5: Comparison: Placebo vs SP 40,000 AUN/ml; Analysis of change from baseline of serum specific IgG4 ATG levels after 10 months (Visit 6); Test type: Superiority; p < 0.001, Mixed Models Analysis; Treatment effect = 2.88, 90% CI 2-sided [2.09 to 3.98]
Statistical Analysis 6: Comparison: Placebo vs SP 80,000 AUN/ml; Analysis of change from baseline of serum specific IgG4 ATG levels after 10 months (Visit 6); Test type: Superiority; p < 0.001, Mixed Models Analysis; Treatment effect = 2.12, 90% CI 2-sided [1.54 to 2.93]
Statistical Analysis 7: Comparison: Placebo vs SP 10,000 AUN/ml; Analysis of change from baseline of serum specific IgG4 AP1 levels after 5 months (Visit 4); Test type: Superiority; p = 0.102, Mixed Models Analysis; Treatment effect = 1.18, 90% CI 2-sided [0.95 to 1.47]
Statistical Analysis 8: Comparison: Placebo vs SP 40,000 AUN/ml; Analysis of change from baseline of serum specific IgG4 AP1 levels after 5 months (Visit 4); Test type: Superiority; p < 0.001, Mixed Models Analysis; Treatment effect = 1.99, 90% CI 2-sided [1.61 to 2.46]
Statistical Analysis 9: Comparison: Placebo vs SP 80,000 AUN/ml; Analysis of change from baseline of serum specific IgG4 AP1 levels after 5 months (Visit 4); Test type: Superiority; p < 0.001, Mixed Models Analysis; Treatment effect = 1.57, 90% CI 2-sided [1.27 to 1.94]
Statistical Analysis 10: Comparison: Placebo vs SP 10,000 AUN/ml; Analysis of change from baseline of serum specific IgG4 AP1 levels after 10 months (Visit 6); Test type: Superiority; p = 0.019, Mixed Models Analysis; Treatment effect = 1.39, 90% CI 2-sided [1.07 to 1.81]
Statistical Analysis 11: Comparison: Placebo vs SP 40,000 AUN/ml; Analysis of change from baseline of serum specific IgG4 AP1 levels after 10 months (Visit 6); Test type: Superiority; p < 0.001, Mixed Models Analysis; Treatment effect = 2.38, 90% CI 2-sided [1.84 to 3.08]
Statistical Analysis 12: Comparison: Placebo vs SP 80,000 AUN/ml; Analysis of change from baseline of serum specific IgG4 AP1 levels after 10 months (Visit 6); Test type: Superiority; p < 0.001, Mixed Models Analysis; Treatment effect = 1.70, 90% CI 2-sided [1.31 to 2.19]
Statistical Analysis 13: Comparison: Placebo vs SP 10,000 AUN/ml; Analysis of change from baseline of serum specific IgG4 AP5 levels after 5 months (Visit 4); Test type: Superiority; p = 0.048, Mixed Models Analysis; Treatment effect = 1.52, 90% CI 2-sided [1.01 to 2.31]
Statistical Analysis 14: Comparison: Placebo vs SP 40,000 AUN/ml; Analysis of change from baseline of serum specific IgG4 AP5 levels after 5 months (Visit 4); Test type: Superiority; p < 0.001, Mixed Models Analysis; Treatment effect = 2.35, 90% CI 2-sided [1.56 to 3.53]
Statistical Analysis 15: Comparison: Placebo vs SP 80,000 AUN/ml; Analysis of change from baseline of serum specific IgG4 AP5 levels after 5 months (Visit 4); Test type: Superiority; p < 0.001, Mixed Models Analysis; Treatment effect = 2.83, 90% CI 2-sided [1.88 to 4.24]
Statistical Analysis 16: Comparison: Placebo vs SP 10,000 AUN/ml; Analysis of change from baseline of serum specific IgG4 AP5 levels after 10 months (Visit 6); Test type: Superiority; p = 0.040, Mixed Models Analysis; Treatment effect = 1.67, 90% CI 2-sided [1.03 to 2.69]
Statistical Analysis 17: Comparison: Placebo vs SP 40,000 AUN/ml; Analysis of change from baseline of serum specific IgG4 AP5 levels after 10 months (Visit 6); Test type: Superiority; p < 0.001, Mixed Models Analysis; Treatment effect = 2.68, 90% CI 2-sided [1.67 to 4.30]
Statistical Analysis 18: Comparison: Placebo vs SP 80,000 AUN/ml; Analysis of change from baseline of serum specific IgG4 AP5 levels after 10 months (Visit 6); Test type: Superiority; p < 0.001, Mixed Models Analysis; Treatment effect = 2.88, 90% CI 2-sided [1.80 to 4.62]

10. Other Pre Specified Outcome: Number and Severity of Local Reactions
Description: The total number and severity (mild, moderate or severe) of local reactions (reported as TEAE) in the active treatment groups and placebo treatment group.
  Intensity grading:
  Mild: Awareness of symptoms but easily tolerated, no disruption of normal activities.
  Moderate: Discomfort enough to cause interference with usual activity. Severe: Incapacitating with inability to work or do usual activity.
Time Frame: Ongoing during 10 months treatment period
Population: The Safety population consists of all randomized subjects who received at least one dose of the study drug. The subjects were included in the treatment group corresponding to the study drug they actually received.
Measure: Number; unit: reactions
Arm/Group | Placebo | SP 10,000 AUN/ml | SP 40,000 AUN/ml | SP 80,000 AUN/ml
Number analyzed (Participants) | 42 | 42 | 42 | 42
reactions
  Total local reactions | 26 | 55 | 91 | 147
  Mild local reactions | 26 | 52 | 82 | 140
  Moderate local reactions | 0 | 3 | 8 | 7
  Severe local reactions | 0 | 0 | 1 | 0

11. Other Pre Specified Outcome: Number and Severity of Systemic Reactions
Description: The total number and severity (Grade I, Grade II or Grade III) of systemic reactions in the active treatment groups and placebo treatment group. The grading was done according to the World Allergy Organization grading system:
  Grade 0: No symptoms or non-immunotherapy-related symptoms Grade I: Mild systemic reactions, symptoms: localized urticaria, rhinitis or mild asthma (PF < 20% decrease from baseline) Grade II: Moderate systemic reactions, symptoms: Slow onset (>15 min) of generalized urticaria and/or moderate asthma (PF < 40% decrease from baseline) Grade III: Severe (non-life-threatening) systemic reactions, symptoms: Rapid onset (<15 min) of generalized urticaria, angioedema or severe asthma (PF > 40% decrease from baseline) Grade IV: Anaphylactic shock, symptoms: Immediate evoked reaction of itching, flushing, erythema, generalized urticaria, stridor (angioedema), immediate asthma, hypotension, etc.
Time Frame: Ongoing during 10 months treatment period
Population: as for outcome 10
Measure: Number; unit: reactions
Arm/Group | Placebo | SP 10,000 AUN/ml | SP 40,000 AUN/ml | SP 80,000 AUN/ml
Number analyzed (Participants) | 42 | 42 | 42 | 42
reactions
  Total Systemic reacions | 69 | 6 | 14 | 27
  Systemic reactions Grade I | 69 | 6 | 14 | 27
  Systemic reactions Grade II | 0 | 0 | 0 | 0
  Systemic reactions Grade III | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event monitoring was performed throughout the conduct of the trial, from subject screening to the end of subject's participation, approximately one year.
Arm/Group | Placebo | SP 10,000 AUN/ml | SP 40,000 AUN/ml | SP 80,000 AUN/ml
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42 | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42 | 1/42 | 0/42 | 1/42
Other Adverse Events (participants affected / at risk) | 26/42 | 36/42 | 33/42 | 36/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=42) | SP 10,000 AUN/ml (N=42) | SP 40,000 AUN/ml (N=42) | SP 80,000 AUN/ml (N=42)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spontaneous abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=42) | SP 10,000 AUN/ml (N=42) | SP 40,000 AUN/ml (N=42) | SP 80,000 AUN/ml (N=42)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 3 (4) | 4 (4) | 9 (11)
Eye pruritus (Eye disorders) | 2 (2) | 1 (1) | 3 (3) | 9 (11)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (4)
Hypoaesthesia oral (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (6) | 4 (5)
Lip pruritus (Gastrointestinal disorders) | 0 (0) | 1 (3) | 3 (4) | 7 (7)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 4 (6) | 2 (2) | 9 (13)
Mouth swelling (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (4) | 7 (10)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (4) | 2 (6) | 4 (5)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 6 (8)
Oral Pruritus (Gastrointestinal disorders) | 3 (7) | 5 (7) | 8 (11) | 11 (14)
Paraesthesia oral (Gastrointestinal disorders) | 3 (5) | 7 (11) | 11 (16) | 11 (17)
Tongue pruritus (Gastrointestinal disorders) | 1 (1) | 3 (3) | 8 (12) | 5 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 13 (18) | 11 (17) | 13 (17) | 10 (14)
Headache (Nervous system disorders) | 11 (17) | 6 (9) | 7 (9) | 11 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (29) | 1 (1) | 2 (2) | 3 (4)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6) | 9 (12) | 13 (16)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No